CLINICAL TRIAL: NCT03316170
Title: Consultation, Advice, and Tailored Support (CATS) for Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jessica Burris (Other)
Collaborators: Kentucky Lung Cancer Research Program (Other)
Responsible Party: Sponsor-Investigator, Jessica Burris, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-17-0495-P3K
Record Dates: First submitted 2017-09-26; First posted 2017-10-20 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Smoking Cessation; Social Stress
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Support + NRT Sampling (Experimental): The treatment group will receive:
  1. a brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs,
  2. a written directory of a range of social support resources delivered via mail,
  3. a brief phone consult (10-15 minutes via phone) germane to smoking cessation,
  4. a written summary of the benefits of smoking cessation, evidence-based approaches to quit, and the basics of nicotine replacement therapy (NRT) delivered via mail, and
  5. a free, 2-week supply of nicotine patches and lozenges delivered via mail.
  Interventions: Behavioral: Social Support; Drug: NRT Sampling
- Social Support (Active Comparator): The control group will receive:
  1. a brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs,
  2. a written directory of a range of social support resources delivered via mail,
  Interventions: Behavioral: Social Support

INTERVENTIONS:
Behavioral: Social Support — A brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs, and a written directory of a range of social support resources delivered via mail.
Drug: NRT Sampling — A brief phone consult (10-15 minutes via phone) germane to smoking cessation akin to "brief advice", a written summary of the benefits of smoking cessation, evidence-based approaches to quit, and the basics of nicotine replacement therapy (NRT) delivered via mail, and a free, 2-week supply of nicotine patches and lozenges delivered via mail.
  Arms: Social Support + NRT Sampling

SUMMARY:
The objectives of this pilot clinical trial are: 1) To evaluate the feasibility and acceptability of a new approach to smoking cessation induction treatment in cancer survivors with low social resources, and 2) To assess the effectiveness of said treatment for key events in the process of smoking cessation.

DETAILED DESCRIPTION:
This is a pilot (Phase II) randomized clinical trial with randomization in a 1:1 ratio. The control group will receive a brief consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs. Additionally, a written directory of a range of social support resources will be delivered to them via mail. The treatment group will receive the aforesaid intervention plus brief advice to quit smoking (10-15 minutes via phone). Additionally, a written summary of the benefits of smoking cessation, evidence-based approaches to quit, and the basics of nicotine replacement therapy (NRT) will be provided via mail. The treatment group will also receive a free, 2-week supply of nicotine patches and lozenges delivered via mail. As a pilot, this study focuses on the outcomes of feasibility (i.e., accrual and retention) and acceptability (e.g., participants' perceptions of appropriateness and effectiveness) as opposed to efficacy (though this is also important). The emphasis on smoking cessation induction (that is, the inducement or promotion of a quit attempt) is an important aspect of the study design and is appropriate for smokers across the continuum of motivation to quit.

ELIGIBILITY:
Inclusion Criteria:

* Cervical or head/neck cancer diagnosis in the past 5 years
* Resident of rural and/or Appalachian Kentucky county at cancer diagnosis
* Current smoker of ≥ 10 cigarettes per day, on average
* Age 18-75 years old
* Able to read, write, and understand English

Exclusion Criteria:

* Unreliable phone access
* Smoking cessation treatment use in past 30 days
* Non-cigarette tobacco use in the past 30 days
* Any FDA contraindication for NRT use, including: allergy to nicotine patches and/or nicotine lozenges; severe kidney or liver disease; unstable angina or serious arrhythmia; epilepsy or seizure disorder; myocardial infarction in the past 3 months
* Cognitive or psychiatric disorder that would interfere with ability to provide informed consent or answer survey questions reliably *

  * Any of these Diagnostic and Statistical Manual-5 (DSM-5) cognitive and psychiatric disorders would make someone ineligible: bipolar; delusional; dissociative; intellectual developmental; neurocognitive; psychotic; schizophreniform, schizophrenia, and schizoaffective.
* For women: breastfeeding, pregnancy, or plan to become pregnant within 6 months
* For women of childbearing potential: unwillingness to use an effective method of birth control (e.g., abstinence, oral contraceptive) while in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Burris, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidani S, Epstein DR, Bootzin RR, Moritz P, Miranda J. Assessment of preferences for treatment: validation of a measure. Res Nurs Health. 2009 Aug;32(4):419-31. doi: 10.1002/nur.20329. PMID 19434647

RESULTS

PARTICIPANT FLOW:
Groups:
- Social Support + NRT Sampling: The treatment group will receive:
  1. a brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs,
  2. a written directory of a range of social support resources delivered via mail,
  3. a brief phone consult (10-15 minutes via phone) germane to smoking cessation,
  4. a written summary of the benefits of smoking cessation, evidence-based approaches to quit, and the basics of nicotine replacement therapy (NRT) delivered via mail, and
  5. a free, 2-week supply of nicotine patches and lozenges delivered via mail.
  Social Support: A brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs, and a written directory of a range of social support resources delivered via mail.
  NRT Sampling: A brief phone consult (10-15 minutes via phone) germane to smoking cessation akin to "brief advice", a written summary of the benefits of smoking cessation, evidence-based approaches to quit, and the basics of nicotine replacement therapy (NRT) delivered via mail, and a free, 2-week supply of nicotine patches and lozenges delivered via mail.
- Social Support: The control group will receive:
  1. a brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs,
  2. a written directory of a range of social support resources delivered via mail,
  Social Support: A brief phone consultation (10-15 minutes via phone) about free or low-cost resources that may help them address unmet social support needs, and a written directory of a range of social support resources delivered via mail.
Period: Overall Study
Arm/Group | Social Support + NRT Sampling | Social Support
Started | 24 | 25
Completed | 17 | 18
Not Completed | 7 | 7
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Population: Each participant is 1 unit in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Support + NRT Sampling | Social Support | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant did not report their age
  years
    number analyzed (Participants) | 23 | 25 | 48
    (all) | 54.78 (9.27) | 56.00 (10.00) | 55.42 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 25 | 49
Distress Thermometer (NCCN) [Mean (Standard Deviation); unit: units on a scale] — The National Comprehensive Cancer Network (NCCN) Distress Thermometer is a single-item measure of overall distress where people respond on a 11-point scale from 0 to 10. Higher scores indicate a worse outcome, as they reflect more distress.
  units on a scale | 4.21 (2.95) | 4.72 (3.45) | 4.47 (3.19)

OUTCOME MEASURES:

1. Primary Outcome: Accrual Percentage
Description: Accrual percentage = (number participants enrolled / number individuals contacted about study participation) multiplied by 100
Time Frame: Day 0 baseline
Population: Across all recruitment methods, a total of 551 individuals were contacted about the study; this number is not tied to study arm. Of these 551 individuals, a subset met the eligibility criteria, enrolled in the study, and were then randomized into one of the study arms.
Measure: Number; unit: percentage of participants enrolled
Groups:
- All Individuals Contacted: All individuals who were contacted about the study.
Arm/Group | All Individuals Contacted
Number analyzed (Participants) | 551
percentage of participants enrolled | 8.9

2. Primary Outcome: Retention
Description: Retention percentage = (number with complete assessments at end of study / number participants enrolled) multiplied by 100
Time Frame: Through study completion, number of assessments at Day 60 follow-up
Population: Participants enrolled in the study
Measure: Number; unit: percentage of participant w/ assessments
Arm/Group | Social Support + NRT Sampling | Social Support
Number analyzed (Participants) | 24 | 25
percentage of participant w/ assessments | 70.8 | 72.0

3. Primary Outcome: Acceptability
Description: Total score on the Treatment Acceptability and Preferences measure (Sidani et al., 2009). This is a 4-item measure with each item scored on a scale from 0 to 4. Total scores are computed as the mean of the 4 individual items, so total scores range from 0 to 4. Higher scores indicate a better outcome, as they reflect greater acceptability of the treatment provided in this clinical trial.
Time Frame: Day 60 follow-up
Population: Analysis based on participants who completed the Day 60 assessment and provided data for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Support + NRT Sampling | Social Support
Number analyzed (Participants) | 16 | 17
score on a scale | 2.84 (1.09) | 1.98 (1.38)
Statistical Analysis 1: Comparison: Social Support + NRT Sampling vs Social Support; Test type: Superiority; p = .06, t-test, 2 sided; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.75 to 0.30], Standard Error of Mean 0.44

ADVERSE EVENTS:
Time Frame: Approximately 2 months
Arm/Group | Social Support + NRT Sampling | Social Support
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 8/24 | 10/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Social Support + NRT Sampling (N=24) | Social Support (N=25)
Breathing difficulty (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Burning in throat or mouth (General disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dizziness (General disorders) | 5 | 8
Dry mouth (General disorders) | 6 | 7
Excessive saliva (General disorders) | 0 | 3
Headache (Nervous system disorders) | 4 | 5
Heartburn (Gastrointestinal disorders) | 4 | 7
Hiccups (Gastrointestinal disorders) | 0 | 3
Insomnia (General disorders) | 7 | 8
Irregular heartbeat (Cardiac disorders) | 2 | 2
Rapid heartbeat (Cardiac disorders) | 2 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 3
Skin itchiness (Skin and subcutaneous tissue disorders) | 2 | 5
Skin redness (Skin and subcutaneous tissue disorders) | 2 | 4
Skin swelling (Skin and subcutaneous tissue disorders) | 1 | 2
Sore mouth (General disorders) | 2 | 4
Sore throat (General disorders) | 4 | 3
Vomiting or nausea (Gastrointestinal disorders) | 1 | 8
Weakness (General disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT03316170/Prot_SAP_000.pdf